CLINICAL TRIAL: NCT05131880
Title: Effectiveness of a Gait Re-education Program on a Sequential Square Treadmill (Tapiz Fisior) in Subjects With Parkison´s Disease
Brief Title: Gait Re-education Program in Subjects With Parkinson´s Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Alberto Bermejo Franco, Principal investigator, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIPI/21/032
Record Dates: First submitted 2021-11-08; First posted 2021-11-23 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'TAPIZ FISIOR' gait re-education program combined with conventional physiotherapy program. (Experimental): The experimental group will undergo a physiotherapy program supplemented by the Fisior Mat Method, with three sessions per week over a 12-week period. Assessments will be conducted at baseline, immediately after the intervention, and at follow-up.
  Interventions: Other: Gait Re-education Program Using the Fisior® Mat Sequential Training System in Subjects with Parkinson's Disease
- Conventional physiotherapy program (Active Comparator): The control group will participate in a physiotherapy program three sessions per week for 12 weeks.
  Interventions: Other: Gait Re-education Program Using the Fisior® Mat Sequential Training System in Subjects with Parkinson's Disease

INTERVENTIONS:
Other: Gait Re-education Program Using the Fisior® Mat Sequential Training System in Subjects with Parkinson's Disease — Randomized controlled study that will include participants diagnosed with Parkinson's disease in mild or moderate stage with altered gait pattern who will be randomized following a simple randomization procedure in which one group will perform an intervention based on a gait re-education program called "TAPIZ FISIOR®"- motor control and learning added to a conventional physiotherapy program; and the other group will perform only a conventional physiotherapy program. The evaluators will be unaware of the patient's treatment condition.

SUMMARY:
Randomized controlled study that will include participants diagnosed with Parkinson's disease in mild or moderate stage with altered gait pattern who will be randomized following a simple randomization procedure in which one group will perform an intervention based on a gait re-education program called "TAPIZ FISIOR"- motor control and learning added to a conventional physiotherapy program; and the other group will perform only a conventional physiotherapy program. The evaluators will be unaware of the patient's treatment status.

DETAILED DESCRIPTION:
All participants interested in participating in the present study will be part of the research project. Once recruited, they will be randomly assigned to two intervention groups: A and B. Group A (control group) will perform a conventional physiotherapy treatment 2/3 sessions per week of 30 minutes duration; on the other hand, group B (intervention group) will perform the treatment of group A and a therapeutic supplement of 2-3 sessions per week of about 30 minutes. During the research period, several measurements of the variables studied will be taken: one before the intervention, one immediately after the end of the intervention, and another measurement 12 weeks after the end of the intervention.

The treatment will be carried out and supervised at all times by qualified physiotherapists, who will explain to you what the treatment consists of, the days you should attend, and the schedules. No adverse effects are expected from this therapy that could pose a risk for health.

ELIGIBILITY:
Inclusion Criteria:

* Older than 50 years.
* Diagnosed Parkinson Disease.
* Not to be institutionalized.
* Barthel index scores of ≥ 60.
* Ability to communicate and to get up and walk at least 10 m (33 ft)

Exclusion Criteria:

* Medical criteria for contraindication of treatment.
* Severe behavioral problems that hinder participation in the training program.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alberto Bermejo Franco, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator: Control Group: Conventional physiotherapy program for Parkinson's disease, designed to address key therapeutic objectives such as improving postural control, increasing gait stability, reducing freezing episodes, enhancing coordination, and minimizing fall risk. The program included gait training to promote step initiation and continuity, balance exercises to improve weight shifting and reactive postural adjustments, stretching to maintain joint mobility and reduce rigidity, and psychomotor activities to enhance proprioception and movement planning. The therapy was conducted by two physiotherapists per center, with sessions lasting 30 minutes, three times per week, over 12 weeks. The pharmacological treatment that participants regularly received was not modified during the intervention to avoid altering the natural progression of the disease.
- Experimental Group: In addition to conventional therapy, the intervention group followed a treatment protocol using the TCS Fisior® sequential square mat, supervised by a trained physiotherapist from each center. This therapy focused on postural control and gait exercises with progressive intensity: low for the first four weeks, moderate until week eight, and high from weeks nine to twelve. Load progression followed a structured protocol, incorporating increased ankle weights, higher repetitions, reduced rest time, and expanded movement directions from anterior to lateral. The effectiveness of this treatment has already shown preliminary evidence in pilot studies conducted on older adults and Parkinson's patients with gait impairments. These additional sessions lasted 30 minutes and were conducted three times per week over the 12-week intervention.
Period: Overall Study
Arm/Group | Active Comparator: Control Group | Experimental Group
Started | 27 | 25
Completed | 27 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: The experimental group will participate in a physiotherapy program with the addition of the Fisior Tapestry Method physiotherapy program, three sessions per week, for 12 weeks.
  An initial assessment will be made at the beginning of the study, another one at the end of the intervention, and another one at follow-up.
  GAIT RE-EDUCATION PROGRAM ON A SEQUENTIAL MAT IN SUBJECTS WITH PARKINSON'S DISEASE: Randomized controlled study that will include participants diagnosed with Parkinson's disease in mild or moderate stage with altered gait pattern who will be randomized following a simple randomization procedure in which one group will perform an intervention based on a gait re-education program called "TAPIZ FISIOR"- motor control and learning added to a conventional physiotherapy program; and the other group will perform only a conventional physiotherapy program. The evaluators will be unaware of the patient's treatment condition.
- Control: The control group will participate in a physiotherapy program three sessions per week for 12 weeks.
  GAIT RE-EDUCATION PROGRAM ON A SEQUENTIAL MAT IN SUBJECTS WITH PARKINSON'S DISEASE: Randomized controlled study that will include participants diagnosed with Parkinson's disease in mild or moderate stage with altered gait pattern who will be randomized following a simple randomization procedure in which one group will perform an intervention based on a gait re-education program called "TAPIZ FISIOR"- motor control and learning added to a conventional physiotherapy program; and the other group will perform only a conventional physiotherapy program. The evaluators will be unaware of the patient's treatment condition.
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.32 (8.39) | 71.37 (7.70) | 71.35 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 15 | 15 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was recorded according to the classification system established by the National Institutes of Health and the United States Office of Management and Budget. Categories include American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, and White. Participants self-reported their race at baseline.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 25 | 27 | 52
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 25 | 27 | 52
Physical Performance: The Short Physical Performance Battery (SPPB) [Mean (Standard Deviation); unit: units on a scale] — The Short Physical Performance Battery (SPPB) assesses lower limb function and mobility through three subtests: standing balance (0-4), 4-m gait speed (0-4), and five-times chair rise (0-4). Subtest scores are summed for a total range of 0-12, with higher scores indicating better performance. The SPPB is widely used to detect mobility limitations, frailty, and disability risk, and has been proposed as an indicator of the mobility subdomain of intrinsic capacity.
  units on a scale | 9.60 (2.47) | 8.78 (2.75) | 9.17 (2.60)
Risk of Falls: FallSkip [Mean (Standard Deviation); unit: units on a scale] — FallSkip is a validated tool for assessing fall risk using a portable inertial sensor placed on the lumbar spine. It evaluates parameters such as balance, gait, reaction time, and strength during standardized tasks. Results are integrated into a global score ranging from 0 (highest risk) to 100 (lowest risk), with higher scores indicating better performance and reduced fall risk.
  units on a scale | 25.4 (13.91) | 26.48 (18.39) | 25.96 (16.08)
Functionality and independence: Barthel Index [Mean (Standard Deviation); unit: units on a scale] — The Barthel Index is a validated scale measuring functionality and independence in activities of daily living (ADLs). It assesses 10 domains including feeding, bathing, dressing, mobility, and continence. Scores range from 0 (total dependence) to 100 (complete independence). Higher scores indicate greater functional autonomy, while lower scores reflect higher dependency and care needs.
  units on a scale | 91.8 (14.13) | 87.59 (12.12) | 89.62 (13.04)

OUTCOME MEASURES:

1. Primary Outcome: Physical Performance: The Short Physical Performance Battery (SPPB)
Description: The Short Physical Performance Battery (SPPB) assesses lower limb function and mobility through three subtests: standing balance (0-4), 4-m gait speed (0-4), and five-times chair rise (0-4). Subtest scores are summed for a total range of 0-12, with higher scores indicating better performance. The SPPB is widely used to detect mobility limitations, frailty, and disability risk, and has been proposed as an indicator of the mobility subdomain of intrinsic capacity.
Time Frame: Before the intervention, up to 15 minutes; and at the end of 12 weeks intervention, up to 15 minutes.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator: Control Group | Experimental Group
Number analyzed (Participants) | 27 | 25
units on a scale
  Pre intervention | 8.78 (2.75) | 9.60 (2.47)
  Post intervention | 8.89 (2.86) | 10.72 (2.01)

2. Primary Outcome: Walk Speed: Timed Up and Go (TUG) Test
Description: The Timed Up and Go (TUG) test assesses basic mobility by measuring the time to stand from a chair, walk three meters, turn, return, and sit down. The time reflects walking speed, balance, turning ability, and overall functional mobility. Shorter times indicate better mobility, while longer times suggest slower gait and potential functional limitations.
Time Frame: Before the intervention, up to 15 minutes; and at the end of 12 weeks intervention, up to 15 minutes.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Active Comparator: Control Group | Experimental Group
Number analyzed (Participants) | 27 | 25
Seconds
  Pre intervention | 0.55 (0.16) | 0.59 (0.13)
  Post intervention | 0.53 (0.19) | 0.67 (0.13)

3. Primary Outcome: Risk of Falls: FallSkip
Description: FallSkip is a validated tool for assessing fall risk using a portable inertial sensor placed on the lumbar spine. It evaluates parameters such as balance, gait, reaction time, and strength during standardized tasks. Results are integrated into a global score ranging from 0 (highest risk) to 100 (lowest risk), with higher scores indicating better performance and reduced fall risk.
Time Frame: Before the intervention, up to 10 minutes; and at the end of 12 weeks intervention, up to 10 minutes.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator: Control Group | Experimental Group
Number analyzed (Participants) | 27 | 25
units on a scale
  Pre intervention | 26.48 (18.39) | 25.4 (13.91)
  Post intervention | 26.85 (16.18) | 21.40 (16.24)

4. Primary Outcome: Functionality and Independence: Barthel Index
Description: The Barthel Index is a validated scale measuring functionality and independence in activities of daily living (ADLs). It assesses 10 domains including feeding, bathing, dressing, mobility, and continence. Scores range from 0 (total dependence) to 100 (complete independence). Higher scores indicate greater functional autonomy, while lower scores reflect higher dependency and care needs.
Time Frame: Before the intervention, up to 20 minutes.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator: Control Group | Experimental Group
Number analyzed (Participants) | 27 | 25
units on a scale | 87.59 (12.12) | 91.8 (14.13)

5. Secondary Outcome: General Satisfaction
Description: The General Satisfaction test is used to assess participants' overall satisfaction with the intervention. Scores range from 0 to 5, where 0 indicates a very poor experience and 5 indicates an excellent experience. The scale reflects the participant's subjective evaluation of the intervention, including factors such as perceived usefulness, comfort, and outcomes. Higher scores represent greater satisfaction. This scale provides a quick and simple way to capture the overall impression of the intervention from the participant's perspective.
Time Frame: At the end of 12 weeks intervention, up to 10 minutes.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator: Control Group | Experimental Group
Number analyzed (Participants) | 27 | 25
units on a scale | 4.3 (0.43) | 4.5 (0.5)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Active Comparator: Control Group | Experimental Group
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 0/27 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-01-31): https://cdn.clinicaltrials.gov/large-docs/80/NCT05131880/Prot_SAP_ICF_000.pdf